CLINICAL TRIAL: NCT05141604
Title: Monocular Visual Confusion for Field Expansion
Brief Title: Feasibility Test of Virtual Reality Obstacle Detection for Low Vision Walking
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Eli Peli, Senior Scientist, Massachusetts Eye and Ear Infirmary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021P003330; R01EY031777 (NIH)
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Hemianopsia; Homonymous Hemianopia; Tunnel Vision; Visual Field Defect, Peripheral; Visual Field Constriction Bilateral; Visual Field Defect Homonymous Bilateral
Keywords: walking; collision; field expansion; visual field loss
MeSH Terms: conditions — Hemianopsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Field expansion view (Experimental): Various configurations of field expansion views will be additionally displayed on HMD
  Interventions: Other: Field expansion view

INTERVENTIONS:
Other: Field expansion view — Overlaid small window on HMD to show the part of the scene in the blind field into portions of the participants' remaining, seeing, field of vision

SUMMARY:
The investigators are developing a new test of pedestrian hazard detection in virtual reality (VR) head-mounted display (HMD) headset, which shows virtual oncoming pedestrians in 3D while subjects are walking in real-world environment, for evaluation of visual field expansion to improve mobility in people with visual field loss.

DETAILED DESCRIPTION:
The investigators will develop a new pedestrian hazard detection test and conduct a single arm interventional clinical trial to evaluate simulated low vision assistive devices in a sample of field loss subjects. Pedestrian detection performance with and without field expansion information will be tested and compared. The study will include 1 to 4 visits (each 2 to 4 hours) depending on the number of trials and experimental conditions (e.g., with and without simulated assistive devices) the subject is comfortable completing. The time between visits may vary depending on scheduling constraints and availability. During each visit, the subject will complete a series of simulated collision avoidance trials in VR requiring the detection and natural avoidance of a colliding pedestrian (alongside non-colliding pedestrians) while physically walking through an empty corridor. The study will be considered minimal-risk since there will be no physical obstacles that present actual collision risks.

ELIGIBILITY:
Inclusion criteria:

* At least 14 years of age (no upper age limit)
* In sufficiently good health to be able to complete sessions lasting 2-3 hours
* Able to understand English
* Able to give voluntary, informed consent
* Able to independently move short distances
* Binocular vision parameters within normal limits (Stereopsis ≤ 100 arc sec on any stereo test)
* Visual field loss, either peripheral field loss (<30 degrees diameter) or hemianopic field loss (blind in half of visual field)
* Better than 20/100 visual acuity in the worse eye

Exclusion criteria:

* Patients with any self-reported physical or mental disabilities, including cognitive dysfunction, balance problems, or other deficits that could impair their ability to respond to the stimuli presented in this study
* Any person with a self-reported medical history (such as pacemaker use or photosensitive epilepsy) or physical condition listed on the device manual of the Oculus / HMD system used for the experiment as a contraindication
* Any self-reported history of seizures (any type) in the last 6 months

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Response time | Through study completion, an average of four months
  During the pedestrian detection task, average response time to the colliding pedestrian with and without prisms

SECONDARY OUTCOMES:
Head movement range | Through study completion, an average of four months
  During the pedestrian detection task, lateral and vertical head movement range to check the head scanning range
Walking speed | Through study completion, an average of four months
  During the pedestrian detection task, the physical walking speed of the subject
Pedestrian detection rate | Through study completion, an average of four months
  Proportion of simulated pedestrians detected (in HMD walking)
Error rate | Through study completion, an average of four months
  Proportion of false alarms and missed targets to total targets

CONTACTS AND LOCATIONS:
Overall Officials: Eli Peli, OD, MSc, Principal Investigator — Senior Scientist
Locations (1):
- Schepens Eye Research Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No